CLINICAL TRIAL: NCT01166399
Title: BOOST: Behavioral Therapy of Obstetric Sphincter Tears: A Cohort Study
Brief Title: Behavioral Therapy Of Obstetric Sphincter Tears
Acronym: BOOST
Status: Completed | Type: Observational
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Office of Research on Women's Health (ORWH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20P01
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence,; bowel incontinence,; pelvic floor disorder
MeSH Terms: conditions — Fecal Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primiparous women with an obstetric anal sphincter tear: Subjects in this trial will be primiparous women who underwent anal sphincter repair at the time of a singleton vaginal delivery. Sphincter tears will be clinically characterized at the time of delivery as <50% tear through the anal sphincter (modified WHO 3a), >50% (modified WHO 3b), or complete tear through the anal sphincter (4th degree). Subjects in this study will not have receive study interventions.

SUMMARY:
The study design will be a cohort study to determine the incidence of FI symptoms at 6, 12 and 24 weeks postpartum in primiparous women sustaining an OASI. At 6, 12 and 24 weeks postpartum, subjects will be contacted by telephone for evaluation of FI symptoms. Symptoms of FI will be defined by at least monthly symptoms of leakage of liquid, solid stool, and mucus. Flatal incontinence will be assessed at 24 weeks, based on the Fecal Incontinence Severity Index, and fecal urgency will be assessed at 24 weeks based on the one question from the Modified Manchester questionnaire. A sample size of approximately 400-450 subjects will be enrolled.

DETAILED DESCRIPTION:
The primary aim of the "BOOST Cohort Study" is to determine the incidence of FI symptoms at 6 and 12 weeks postpartum in primiparous women sustaining an OASI.

Secondary aims of the cohort study are:

1. To determine the incidence rates of FI symptoms at 24 weeks post delivery in primiparous women sustaining an OASI
2. To examine the relationship between the modified WHO sphincter tear classification types and FI symptoms
3. To examine predictors (socio-demographic, physical and clinical) associated with WHO sphincter tear classifications (3a, 3b and 4) and predictors associated with FI symptoms
4. To evaluate the incidence of fecal urgency and flatal incontinence at 24 weeks postpartum in primiparous women sustaining an OASI.

ELIGIBILITY:
Inclusion Criteria Assessed by 2 weeks postpartum

1. Vaginal delivery >= 28 weeks singleton gestation
2. Documented repair to the anal sphincter at delivery
3. First vaginal delivery
4. Ambulatory
5. Able to give informed consent 6 Adult women >= 18 years of age

Inclusion Criteria at 2 weeks postpartum

1. Inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease)
2. Pre-pregnancy ano-rectal surgery (e.g., surgery for hemorrhoids, fissures, sphincterotomy)
3. Pre-pregnancy FI (defined as the leakage of liquid/solid stool and mucus >= once per month for at least 12 weeks prior to this pregnancy)
4. Neurological condition that would predispose to FI (e.g., spinal cord injury, multiple sclerosis)
5. Presence of rectovaginal fistula
6. Any participation in other pharmacologic or behavioral studies for FI
7. Previous pregnancy >=28 weeks delivered vaginally or by Cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in this trial will be primiparous women who underwent anal sphincter repair at the time of a singleton vaginal delivery. Sphincter tears will be clinically characterized at the time of delivery as <50% tear through the anal sphincter (modified WHO 3a), >50% (modified WHO 3b), or complete tear through the anal sphincter (4th degree).
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of FI | 6 and 12 months postpartum
  The primary aim for this study is to determine the incidence of FI symptoms (based on the FISI)at 6 and 12 weeks postpartum in primiparous women sustaining an OASI.

SECONDARY OUTCOMES:
Incidence of FI | 24 weeks postpartum
  A secondary aim for this study is to determine the incidence of FI symptoms (based on the FISI) at 24 weeks postpartum in primiparous women sustaining an OASI.
Fecal urgency | 24 weeks postpartum
  Fecal urgency will be assessed at 24 weeks based on the one question from the Modified Manchester questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Holly E Richter, PhD, MD, Study Chair — University of Alabama at Birmingham
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Loyola University, Maywood, Illinois
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Richter HE, Nager CW, Burgio KL, Whitworth R, Weidner AC, Schaffer J, Zyczynski HM, Norton P, Jelovsek JE, Meikle SF, Spino C, Gantz M, Graziano S, Brubaker L; NICHD Pelvic Floor Disorders Network. Incidence and Predictors of Anal Incontinence After Obstetric Anal Sphincter Injury in Primiparous Women. Female Pelvic Med Reconstr Surg. 2015 Jul-Aug;21(4):182-9. doi: 10.1097/SPV.0000000000000160. PMID 25679358